GALDERMA
Title
43USSA1705 Sculptra Clinical Study Protocol

MA-37876

Print date:

2022-07-26 17:40

# A randomized, evaluator-blinded, multi-center study to evaluate the safety and effectiveness of Sculptra Aesthetic for correction of nasolabial folds

Study product: Sculptra® Aesthetic

Clinical trial number (CTN): 43USSA1705

Sponsor: Q-Med AB, a Nestle Skin Health Affiliate





Doc id 43USSA1705 Sculptra Clinical Study Protocol ♣ GALDERMA **MA-37876** 

Print date:

2022-07-26 17:40

## **Study Administrative Structure**



Further details on all participating Investigators and the complete administrative structure of the study are found in the study files. Note that administrative changes are to be documented in the study files without requiring a Clinical Investigational Plan (CIP) amendment.

Doc id 43USSA1705 Sculptra Clinical Study Protocol ♣ GALDERMA MA-37876

Print date:

2022-07-26 17:40

# **Sponsor Signatures**

The CIP is electronically signed in the document management system within the Q-Med AB quality management system by the representatives listed below.



Doc id 43USSA1705 Sculptra Clinical Study Protocol GALDERMA MA-37876

Print date:

2022-07-26 17:40

# Synopsis

| Title of study | A randomized, evaluator-blinded, multi-center study to evaluate the safety and effectiveness of Sculptra Aesthetic for correction of nasolabial folds |
|---|---|
| Clinical Trial<br>Number | 43USSA1705 |
| Countries involved | United States |
| Number of sites | Approximately 5 sites |
| Number of subjects | Approximately 80 total subjects will be enrolled in the study |
| Target<br>Indication | Sculptra Aesthetic is indicated for use in immune competent people as single regimen for correction of shallow to deep nasolabial fold contour deficiencies and other facial wrinkles. The development proposed is within the approved indication to assess the safety and effectiveness after changes in reconstitution and injection procedures. |
| Safety Objective<br>and Endpoints | The objective is to evaluate the safety of Sculptra Aesthetic as a single regimen for correction of Nasolabial Fold (NLF) contour deficiencies after changes in reconstitution and injection procedures compared to the approved label. Safety endpoints Incidence, intensity, time to onset and duration of adverse events collected throughout the study period. |
| | Incidence, intensity, time to onset and number of days of pre-<br>defined expected post-treatment events collected using subject |

Doc id 43USSA1705 Sculptra Clinical Study Protocol . GALDERMA MA-37876

Print date:

2022-07-26 17:40

| | diaries for 28 days from each treatment. |
|---|---|
| Effectiveness<br>Objectives and<br>Endpoints | The objective is to evaluate the effectiveness of Sculptra Aesthetic as a single regimen for correction of NLF contour deficiencies after changes in reconstitution and injection procedures compared to the approved label. |
| | Primary effectiveness endpoint |
| | Change from baseline on both sides of the face as assessed by the Blinded Evaluator using at 48 Weeks after the first treatment session. |
| Study Design | This is a prospective, randomized, evaluator-blinded, multicenter US |
| Study Design | study. |
| Subject<br>Participation | A subject may be involved in the study for approximately 52 weeks from screening to the final follow-up visit. |
| Enrollment | Written informed consent will be obtained before any study related procedures is performed. Subjects will be screened for eligibility within 30 days prior to injection. The screening visit and baseline visit may be performed on the same day. Subsequent to screening, eligible subjects will be randomized in the study. |
| | This study will include at least eight (8) subjects with Fitzpatrick Skin Type (FST) IV and at least eight (8) subjects with FST V-VI. |

43USSA1705 Sculptra Clinical Study Protocol

-----

Doc id

MA-37876

# Inclusion criteria

Effective date: 2019-02-21 18:33

The subjects must meet the following criteria to be eligible for the study:

- 1. Subjects willing to comply with the requirements of the study and providing a signed written informed consent.
- 2. Immune-competent men or women over 21 years of age







# Exclusion criteria

The presence of any of the following exclusion criteria will exclude a subject from enrollment in the study:

- 1. Known/previous allergy or hypersensitivity to any of the Sculptra Aesthetic constituents.
- Known/previous allergy or hypersensitivity to lidocaine and other local anesthetics, e.g. amide-type anesthetics, or topical anesthetics or nerve blocking agents.
- Previous or present multiple allergies or severe allergies, such as manifested by anaphylaxis or angioedema, or family history of these conditions.

4.

Print date: 2022-07-26 17:40

GALDERMA
Title
43USSA1705 Sculptra Clinical Study Protocol

MA-37876

Effective date: 2019-02-21 18:33




Effective date: 2019-02-21 18:33

43USSA1705 Sculptra Clinical Study Protocol

**MA-37876** 

Doc id



Doc id 43USSA1705 Sculptra Clinical Study Protocol GALDERMA **MA-37876** 



Doc id 43USSA1705 Sculptra Clinical Study Protocol GALDERMA MA-37876

Print date:

2022-07-26 17:40



Doc id 43USSA1705 Sculptra Clinical Study Protocol ♣ GALDERMA **MA-37876** 



Effective date: 2019-02-21 18:33

Title
43USSA1705 Sculptra Clinical Study Protocol

Doc id

Print date:

MA-37876

2022-07-26 17:40





Print date:

2022-07-26 17:40



Doc id 43USSA1705 Sculptra Clinical Study Protocol ♣ GALDERMA **MA-37876** 

### **Abbreviations and Definitions of Terms**

AE Adverse event

**AESI** Adverse event of special interest

Blinded Evaluator An evaluator responsible for independent evaluation of treatment

result(s). The evaluator must not be involved in the treatment of the

Print date:

2022-07-26 17:40

subject.

CE French: Conformité Européenne **CFR** Code of Federal Regulations

Childbearing potential A female (including pre-menopausal subjects) capable of becoming

> pregnant. This includes women on oral, injectable or mechanical contraception; women who are single, women whose husbands have been vasectomized or whose husbands have received or utilizing

mechanical contraceptive devices.

CIP Clinical Investigational Plan

**CRF** Case report form

**CRO** Contract research organization

**CTA** Clinical trial agreement **CTN** Clinical trial number CV Curriculum vitae

Device deficiency Inadequacy of a medical device with respect to its identity, quality,

durability, reliability, safety or performance (includes malfunctions,

use errors, and inadequate labelling)

**DMP** Data management plan **eCRF** Electronic case report form

ET **Early Termination** 

**FDA** United States Food and Drug Administration

First treatment Initial injection of study product

**FST** Fitzpatrick Skin Type

G Gauge

Good Clinical Practice **GCP** 

HA Hyaluronic acid

**HIPAA** Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

Informed Consent Form **ICF** 

International Conference on Harmonisation **ICH** 

**IFU** Instructions for use

Doc id 43USSA1705 Sculptra Clinical Study Protocol ♣ GALDERMA **MA-37876** 

Investigational product Medical device being assessed for safety or performance in a study.

"Investigational product" is the same as "study device",

"investigational device", or "investigational medical device"

Institution Any public or private entity or agency or medical or dental facility

where a clinical study is conducted.

Investigator The Principal Investigator (PI) or other qualified person, i.e. sub-

> investigator, designated and supervised by the PI at a study site to perform critical study-related procedures or to make important study-related decisions as specified on the signature and delegation

Print date:

2022-07-26 17:40

Investigator file Essential documents relating to a clinical study as defined in

applicable GCP guidance document and maintained by the

Investigator.

ΙP **Investigational Product IPL** Intense Pulsed Light

**IRB** Institutional Review Board

ISO International Organization for Standardization

Intrauterine Device **IUD** 

MedDRA Medical dictionary for regulatory activities

Nasolabial Fold (NLF) Lines between the nose and the corner of the mouth

**NSAID** Non-Steroidal Anti-Inflammatory

Drugs

**PLLA** Poly-L-lactic acid

ΡI Principal Investigator; qualified person responsible for conducting

the study at a study site

PP Per Protocol PT Preferred Term QA Quality Assurance RARegulatory Authority

**ROPI** Report of Prior Investigations, i.e. compilation of the current

clinical and non-clinical information on the investigational product,

relevant to the clinical study

Reference product Sculptra Aesthetic reconstituted with 5 mL of SWFI

Serious Adverse Event SAE **SDV** Source Data Verification **SWFI** Sterile Water for Injection

SOC System Organ Class SOE Schedule of Events

| GALDERMA Title 43USSA1705 Sculptra Clinical Study Protocol | Doc id MA-37876 |
|---|---|
|---|---|

Print date:

2022-07-26 17:40

Sponsor file

Essential documents relating to a clinical study as defined in applicable GCP guidance document and maintained by the Sponsor.

Study files

The Investigator file and the Sponsor file

Study products

The investigational products and the reference product under study

Study site

UPT

Urine Pregnancy Test

WHO World Health Organization



Title
43USSA1705 Sculptra Clinical Study Protocol

Doc id

MA-37876

# **Table of Contents**

| Stud | ly Admir | nistrative Structure | 2 |
|---|---|---|---|
| Spor | nsor Sign | natures | 3 |
| Syno | opsis | | 4 |
| Abb | reviation | ns and Definitions of Terms | 14 |
| List | of Table | S | 20 |
| List | of Figur | es | 20 |
| 1. | C | Considerations | |
| 1. | 1.1 | Statement of ethical compliance | |
| | 1.2 | Application to Institutional Review Board and/or Regulatory Authorities | |
| 2. | Backer | ound Information | |
| _, | 2.1 | Indication and population description. | |
| | 2.2 | Investigational and Reference product description | |
| | 2.3 | Clinical documentation | |
| | 2.4 | Study rationale and justification for design | 23 |
| | 2.5 | Risks and benefits | 24 |
| 3. | Objecti | ives and Endpoints | 25 |
| | 3.1 | Safety objective and endpoints | 25 |
| | 3.2 | Effectiveness objective and endpoints | 26 |
| 4. | Design | of the Study | 26 |
| | 4.1 | General outline | 26 |
| | 4.2 | Number of subjects | 29 |
| | 4.3 | Duration of subject participation | 29 |
| | 4.4 | Randomization and blinding | 29 |
| | 4.5 | Medical history | 30 |
| | 4.6 | Prior and concomitant therapies | 30 |
| | 4.6.1 | Definition | |
| | 4.6.2 | Concomitant therapies are defined as follows: | |
| | 4.6.3 | Concomitant medication, treatments and procedures | |
| | 4.7 | Schedule of events | 32 |

Print date:

2022-07-26 17:40

| | <u> </u> | P. Committee of the Com | |
|---|---|---|---|
| 5. | Subjects | S | |
| | 5.1 | Subject information and informed consent | |
| | 5.2 | Inclusion criteria | |
| | 5.3 | Exclusion criteria | |
| | 5.4 | Screening and subject number | |
| | 5.5 | Withdrawal of subjects | 44 |
| 6. | Study Pr | roducts | 45 |
| | 6.1 | Investigational product | 45 |
| | 6.2 | Reference product | 45 |
| | 6.3 | Additional study supplies | 45 |
| | 6.4 | Packaging, labeling, and storage | 46 |
| | 6.5 | Product accountability | 46 |
| | 6.6 | Treatment | 47 |
| | 6.6.1 | Treatment procedure | 47 |
| | 6.6.2 | Treatment regimen | 47 |
| | 6.6.3 | Post injection care | 48 |
| | 6.6.4 | Post treatment care | 48 |
| | 6.6.5 | Post trial provisions | 48 |
| 7. | Safety A | Assessments | 49 |
| | 7.1 Assess | sment of AEs by direct questioning to subject and evaluation of subject | 49 |
| | 7.6 | Laboratory assessments | 50 |
| | 7.7 | Adverse events | 51 |
| | 7.7.1 | Definition of an adverse event | 51 |
| | 7.7.2 | Definition of a serious adverse event | 51 |
| | 7.7.3 | Recording instructions | 51 |
| | 7.7.3.1 | Intensity | 52 |
| | 7.7.3.2 | Causal relationship and seriousness | 52 |
| | 7.7.4 | Reporting of adverse events | 53 |
| | 7.7.6 | Reporting of serious adverse events | 53 |
| | 7.7.7 | Stopping Rule | |

| ♣ GALDERMA | 43USSA1705 Sculpt |
|------------|-------------------|
|------------|-------------------|

| 1 ILIC | | | | |
|-------------|----------|----------|-------|----------|
| 3USSA1705 S | Sculptra | Clinical | Study | Protocol |

Doc id

# **MA-37876**

| | 7.7.9 | Pregnancy | 55 |
|---|---|---|---|
| | 7.7.10 | Anticipated adverse events | 56 |
| | 7.8 | Device deficiencies | 56 |
| | 7.8.1 | Definition of a device deficiency | 56 |
| | 7.8.2 | Recording instructions | 56 |
| | 7.8.3 | Reporting of device deficiencies | 56 |
| 8. E | ffective | ness Assessments | 57 |
| 9 | Data H | Iandling and Management | 60 |
| | 9.1 | Data management | |
| | 9.2 | Electronic case report forms | 60 |
| | 9.2.1 | Data entry | 61 |
| | 9.2.2 | The query process | 61 |
| | 9.2.3 | User identification | 61 |
| | 9.2.4 | Audit trail | 61 |
| | | rce documents | |
| | | ord keeping and access to source data | |
| | 9.5 Doc | ument and data retention | 62 |
| 10 | Statisti | ical Methods | 62 |
| | 10.1 Ge | eneral | 62 |
| | 10.2 An | alysis populations | 63 |
| | 10.3 | Demographics, baseline assessments, and subject characteristics | 63 |
| | 10.4 Pri | mary effectiveness analysis | 63 |
| | 10.5 Sec | condary effectiveness analysis | 64 |
| | 10.6 | Safety analysis | |
| | 10.7 | Subgroup analyses | 65 |
| | 10.8 | Handling of missing data | |
| | 10.9 | Interim analysis | |
| | 10.10 | Withdrawals and deviations | |
| | 10.11 | Sample size | 65 |
| 11 | Protect | tion of personal data | 66 |
| 12 | Quality | y Control and Quality Assurance | 66 |
| | 12.1 | Quality control | 66 |
| | 12.2 | Quality assurance | 67 |
| | 12.3 | Changes to the clinical study protocol | 67 |
| 13 | Financ | ring, Indemnification, and Insurance | 67 |
| 14 | Publica | ation Policy | 67 |

| | | | Print date: | 2022-07-26 17:40 |
|---|---|---|---|---|
| GAL | DERMA | Title 43USSA1705 Sculptra Clinical Study Protocol | Doc id MA-3 | 37876 |
| 15 | Suspensio | on or Premature Termination | | 68 |
| 16 | | ·s | | |
| 17 | Appendic | es | | 70 |
| Li | ist of Tal | oles | | |
| | ist of Fig | ures<br>pendices | | |
| | 10 | | | |



Print date:

2022-07-26 17:40

### 1. Ethical Considerations

### 1.1 Statement of ethical compliance

The study shall be conducted in compliance with the Clinical Trial Agreement (CTA), the Clinical Investigational Plan (CIP), Good Clinical Practice (GCP), and applicable regional or national regulations. The study shall be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki<sup>1</sup>.

The study shall follow the international standard for clinical study of medical devices for human subjects, ISO14155 as applicable for US regulations and the International Conference on Harmonization (ICH) guideline for GCP (E6) as applicable for medical device.

### 1.2 Application to Institutional Review Board and/or Regulatory Authorities

It is the responsibility of the Principal Investigator (PI) to obtain approval of the CIP/CIP amendment from the Institutional Review Board (IRB). The study shall not begin until the required favorable opinion from the IRB has been obtained. The PI shall file all correspondence with the IRB in the Investigator file and copies of IRB approvals shall be forwarded to the Sponsor. Any additional requirements imposed by the IRB or regulatory authorities (RA), shall be followed.

The study requires application for approval from the US Food and Drug Administration (FDA). The study will not be started until the Sponsor has received written approval or until the statutory waiting period from the appropriate authority has elapsed.

The collection, access to, processing, and transfer of protected health information or sensitive personal data shall be carried out in accordance with applicable regional or national regulations.

### 2. Background Information

### 2.1 Indication and population description



Effective date: 2019-02-21 18:33

Title
43USSA1705 Sculptra Clinical Study Protocol

Doc id

Print date:

MA-37876

2022-07-26 17:40

2.2 Investigational and Reference product description



Effective date: 2019-02-21 18:33

Title
43USSA1705 Sculptra Clinical Study Protocol

Doc id

Print date:

**MA-37876** 

2022-07-26 17:40



2.3 Clinical documentation



2.4 Study rationale and justification for design



Print date: Doc id 43USSA1705 Sculptra Clinical Study Protocol ♣ GALDERMA MA-37876

2022-07-26 17:40





Doc id 43USSA1705 Sculptra Clinical Study Protocol GALDERMA MA-37876

Print date:

2022-07-26 17:40



## **Objectives and Endpoints**

### Safety objective and endpoints

### Safety objective

The objective is to evaluate the safety of Sculptra Aesthetic as a single regimen for correction of NLF contour deficiencies after changes in reconstitution and injection procedures compared to the approved label.

### Safety endpoints

- Incidence, intensity, time to onset and duration of adverse events collected throughout the study period.
- Incidence, intensity, time to onset and number of days of pre-defined expected posttreatment events collected using subject diaries for 28 days from each treatment.



Doc id 43USSA1705 Sculptra Clinical Study Protocol GALDERMA MA-37876

Print date:

2022-07-26 17:40

#### 3.2 Effectiveness objective and endpoints

### Effectiveness objective

The objective is to evaluate the effectiveness of Sculptra Aesthetic as a single regimen for correction of NLF contour deficiencies

### Primary effectiveness endpoint

Change from baseline on both sides of the face as assessed by the Blinded Evaluator at 48 Weeks after the first treatment session. using



## **Design of the Study**

#### 4.1 General outline

This is a 48-week, randomized, evaluator-blinded, parallel-group, multi-center, study to evaluate the safety and effectiveness of treatment with Sculptra Aesthetic for correction of NLF contour deficiencies after changes in reconstitution and injection procedures compared to the approved label.

Approximately 64 subjects requiring correction of NLFs will be enrolled and randomized in a 2:1 ratio to treatment with Sculptra Aesthetic reconstituted with 8 mL of SWFI (treatment group) or to Sculptra Aesthetic reconstituted with 5 mL of SWFI (reference group). In addition, eight (8) subjects with FST IV and eight (8) subjects with FST V-VI will be included but not randomized. These subjects will be treated with Sculptra Aesthetic reconstituted with 8 mL of SWFI. When these numbers of FST IV-VI have been treated, any additional FST IV-VI will be randomized in a 2:1 ratio (8 mL:5 mL).

Approximately 60 subjects will be treated with Sculptra Aesthetic reconstituted with 8 mL of SWFI and a reference group of approximately 20 subjects will be treated with Sculptra Aesthetic reconstituted with 5 mL of SWFI as according to the current label.



Investigator blinding will be accomplished by using a Treating Investigator to administer the

GALDERMA
Title
43USSA1705 Sculptra Clinical Study Protocol

MA-37876

Print date:

2022-07-26 17:40

treatments and a Blinded Evaluator, to whom randomization and treatment are concealed, to conduct the blinded assessments. In addition, the Blinded Evaluator should not be allowed to retrieve study supplies or be present during the opening of the study supplies or injection procedure. All documents with information regarding study products and randomization assignment should be kept in a separate binder not available to the blinded evaluator. Safety assessments will be performed by non-blinded personnel.

Eligible subjects randomized to receive treatment will be injected by the Treating Investigator at Day 1. The method of injection is at the discretion of the treating Investigator according to Sections 2.2 and 6.6.

Sufficient amount of product should be injected to achieve optimal correction of the NLFs, in the opinion of the Treating Investigator and subject.





| • CALDEDAAA | 43USSA1705 Sculptra Clinical Study Protocol | Doc id |
|-------------|---------------------------------------------|----------|
| GALDERMA | | MA-37876 |

Print date:

2022-07-26 17:40

#### 4.2 Number of subjects

Approximately 80 subjects will be recruited at approximately 5 sites in the USA.

The duration of enrollment is expected to be approximately 3 months.

#### **Duration of subject participation** 4.3

A subject may be involved in the study for approximately 52 weeks from screening to the final follow-up visit.

End of study is when enrollment has reached the target number of subjects and all subjects have completed the last study visit.

### Randomization and blinding



#### 4.4.2 Blinding

Blinding will be accomplished by using a Treating Investigator to administer the treatments and a Blinded Evaluator, to whom randomization and treatment are concealed, to conduct the blinded assessments. The Treating Investigator will <u>not</u> be blinded. The Blinded Evaluator is not allowed to discuss treatments with the Treating Investigator or subjects. No study related documents that contain information regarding the treatment of subjects should be available to the Blinded Evaluator. Safety assessments will be performed by non-blinded personnel who are qualified by training and experience.

### 4.4.3 Emergency Unblinding

Not applicable as the Treating Investigator is unblinded.



### 4.5 Medical history

History of surgical events and medical conditions should be documented (including any prior dermatological procedures or implants) in the source and electronic case report forms (eCRF) using medical terminology.

### 4.6 Prior and concomitant therapies

### 4.6.1 Definition

Therapies are defined as medications, treatments and procedures.

Prior therapies are defined as therapies that have been stopped within 30 days of the Screening visit or within the timelines specified in the Inclusion/Exclusion criteria. Prior therapies as defined above are to be recorded in source documents and the eCRF.

### 4.6.2 Concomitant therapies are defined as follows:

- 1. Any therapy ongoing at the time of the Screening visit,
- Any changes to existing therapies (such as changes in dose or formulation) during the course of the study, or
- 3. Any new therapies started after the Screening visit.

### 4.6.3 Concomitant medication, treatments and procedures

Except as noted below, concomitant medications or other treatments or procedures may be utilized when the Investigator or his/her authorized designee considers it medically necessary.

Information regarding any use of concomitant medications, including prescription and over- the-counter medications administered during the study is to be recorded in source documents and the eCRF. The generic name or the trade name of all concomitant medication or a description of the procedure and the reason for its use shall also be documented accordingly.

The following medications, treatments, and procedures are restricted or prohibited during the study:





If a treated subject has used any of the above prohibited medications or procedures, the subject should, for safety reasons, continue in the study for the scheduled follow-up visits. Before any further study treatments are provided, the Treating Investigator should discuss the subject with the Medical Monitor.

Print date: 2022-07-26 17:40

GALDERMA

Title
43USSA1705 Sculptra Clinical Study Protocol

MA-37876

Doc id

Numeric Pain Scale (NPS)  $X^{7,2}$ X7,2 X7,2

**Effective** 

Effective date: 2019-02-21 18:33


Effective date: 2019-02-21 18:33












Effective date: 2019-02-21 18:33

Print date:

2022-07-26 17:40

Doc id 43USSA1705 Sculptra Clinical Study Protocol ♣ GALDERMA MA-37876 ne 

Effective date: 2019-02-21 18:33

Print date:

2022-07-26 17:40





2022-07-26 17:40

## Subjects

### Subject information and informed consent

The Investigator or his/her authorized designee must always use the IRB-approved subject information and informed consent form (ICF) and it must not be changed without prior discussion with the Sponsor and approval from the applicable IRB.

It is the responsibility of the Investigator or his/her authorized designee to give each subject, prior to inclusion in the study, full and adequate verbal and written information regarding all aspects of the clinical study that are relevant to the subject's decision to participate throughout the study, e.g. explain the purpose and procedures of the study, the duration and number of expected participants, possible risks involved, and the opinion of the IRB. The subject shall be informed that the participation is confidential and voluntary and that the subject has the right to withdraw from the study at any time, without any effect on his/her future medical care, treatment or benefits to which the subject is otherwise entitled. The information shall be provided in a language clearly and fully understandable to the subject. The subject shall be given sufficient time to read and understand the informed consent form and to consider participation in the study. Before any study-related activities are performed, the informed consent form shall be personally signed and dated by the subject and the Investigator or his/her authorized designee responsible for conducting the informed consent process.

All original signed informed consent forms shall be filed in the Investigator file. The subject shall be provided with a copy of the signed and dated informed consent form and any other written information.

The Investigator shall ensure that important new information is provided to new and existing subjects throughout the study.

#### Inclusion criteria

The subjects must meet the following criteria to be eligible for the study:

- 1. Subjects willing to comply with the requirements of the study and providing a signed written informed consent.
- Immune-competent men or women over 21 years of age



Print date:

2022-07-26 17:40



#### 5.3 Exclusion criteria

The presence of any of the following exclusion criteria will exclude a subject from enrollment in the study:

- 1. Known/previous allergy or hypersensitivity to any of the Sculptra Aesthetic constituents.
- 2. Known/previous allergy or hypersensitivity to lidocaine and other local anesthetics, e.g. amide-type anesthetics, or topical anesthetics or nerve blocking agents.
- 3. Previous or present multiple allergies or severe allergies, such as manifested by anaphylaxis or angioedema, or family history of these conditions.



♣ GALDERMA

Effective date: 2019-02-21 18:33

43USSA1705 Sculptra Clinical Study Protocol

**MA-37876** 

Doc id





2022-07-26 17:40

#### 5.4 Screening and subject number

Prior to any study procedures being conducted, the subject must sign the informed consent form. Each subject who has signed the informed consent form will be assigned a subject number. The subject number, subject name, and other information sufficient to link the eCRF to the medical records (e.g. national identification number, chart number, etc.) shall be recorded.

A screen failure is a subject who signed the informed consent but never enrolled (i.e. was randomized and/or received treatment) in the study. For screen failures, the subject's source documents should indicate which assessments have been made and the reason why the subject was determined to be a screen failure. A subject is considered enrolled when they have signed the ICF and are randomized and/or treated.

During the study conduct, the Blinded Evaluators should not have access to any subject's source documents that identify the subject.

#### 5.5 Withdrawal of subjects

Each subject shall be advised in the informed consent form that the subject has the right to withdraw from the study at any time, for any reason, without prejudice. Subjects may also be discontinued from this study if the Investigator determines that it is in the subject's best interest to do so, and may be withdrawn at the Investigator's discretion at any time.



The reason and date for withdrawal shall be documented in the eCRF. When possible, an explanatory comment shall be added to further explain the reason for withdrawal. If withdrawal of a subject occurs during a regular study visit, the eCRF for that specific visit shall be completed as far as possible.



2022-07-26 17:40

If withdrawal of a subject occurs between regular study visits, the subject should when possible (irrespective of the reason for withdrawal) be scheduled for a termination visit to document subject outcome for the secondary endpoints.

If a subject is withdrawn from the study, all data collected until the time of withdrawal will be used in the analyses.

Subjects who receive product and are withdrawn or discontinued from the study will not be replaced.

For AEs still ongoing at the time of withdrawal, see Section 7.7.8.

## **Study Products**

The term "study product" refers to Sculptra Aesthetic (i.e. the investigational product and the reference product). The study product will be provided by the sponsor.

#### Investigational product 6.1

Sculptra Aesthetic is an injectable implant containing microparticles of poly-L-lactic acid (PLLA), carboxymethylcellulose, non-pyrogenic mannitol and sterile water for injection (SWFI). Sculptra Aesthetic is available in 367.5 mg dose vials and is to be reconstituted prior to use by the addition of 8 mL SWFI to form a sterile non-pyrogenic suspension.

#### 6.2 Reference product

Sculptra Aesthetic is an injectable implant containing microparticles of PLLA, carboxymethylcellulose, non-pyrogenic mannitol and SWFI. Sculptra Aesthetic is available in 367.5 mg dose vials and is to be reconstituted prior to use by the addition of 5 mL SWFI to form a sterile non-pyrogenic suspension.





2022-07-26 17:40



#### Product accountability

The study products will be released to the Investigator or his/her authorized designee after study approvals have been received from the FDA and IRB and the CTA has been signed by all parties.

The Investigator must ensure that the study products are kept in a secure location, with access limited to those authorized by the Investigator.

The study products must be traceable from the manufacturer to their use in subjects until return or disposal. It is therefore important that the Investigator maintains accurate product accountability records, i.e. documentation of the physical location of all investigational products, deliveries, and return of investigational products between the Sponsor and the Investigator, and documentation of administration of product to the subject.

When the study is completed, all unused or expired investigational product at each study site shall be returned to the Sponsor representative for destruction, or be destroyed locally at the site if documented as agreed with Sponsor.

Any malfunctioning investigational products shall be reported as described in Section 7.8.

Products deliberately or accidentally destroyed during shipment or at a study site shall be accounted for and documented. Used vials, syringes, needles, and any unused material must be discarded immediately after the treatment session and must not be reused due to risk for contamination of the unused material and the associated risks including infections according to standard procedures at the site. Disposal of hazardous material, i.e. syringes and needles must conform to applicable laws and regulations.

The study products must not be used outside of the study.

All study products sent to the Investigator will be accounted for and no unauthorized use is permitted.

Effective date: 2019-02-21 18:33

Title
43USSA1705 Sculptra Clinical Study Protocol

Doc id

Print date:

**MA-37876** 

2022-07-26 17:40





♣ GALDERMA

Effective date: 2019-02-21 18:33

Title
43USSA1705 Sculptra Clinical Study Protocol

Doc id

Print date:

**MA-37876** 

2022-07-26 17:40



Effective date: 2019-02-21 18:33

Title
43USSA1705 Sculptra Clinical Study Protocol

Doc id

Print date:

**MA-37876** 

2022-07-26 17:40

# 7. Safety Assessments

7.1 Assessment of AEs by direct questioning to subject and evaluation of subject





Doc id 43USSA1705 Sculptra Clinical Study Protocol ♣ GALDERMA **MA-37876** 

Print date:

2022-07-26 17:40

#### 7.7 Adverse events

#### Definition of an adverse event

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons<sup>7</sup>, whether or not related to the study product.

This definition includes:

- events related to the investigational product or the reference product a)
- b) events related to the procedures involved

#### Definition of a serious adverse event

A serious adverse event (SAE) is an AE that:

- a) led to death,
- b) led to serious deterioration in the health of the subject, that either resulted in
  - 1. a life-threatening<sup>8</sup> illness or injury, or
  - 2. a permanent impairment of a body structure or body function, or
  - 3. in-patient or prolonged hospitalization<sup>9</sup>, or
  - 4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
- c) led to fetal distress, fetal death, or a congenital abnormality or birth defect

An AE does not need to be recorded as a SAE if it only represents a relapse or an expected change or progression of the condition that was the cause of the treatment, without the development of new symptoms and signs.

In cases of doubt, whether an AE fulfils a serious criterion or not, there should be a predisposition to report as a SAE rather than not report as such (see Section 7.7.6).

#### Recording instructions 7.7.3

Each subject with an AE occurring after enrollment through study exit should be fully recorded in the source document(s) for further transcription to the eCRF. Each subject should be questioned about AEs at each study visit following randomization and or treatment. The question asked should be: "Since your last clinical visit have you had any health problems?" Information on AEs can also be obtained from signs and symptoms detected during each examination.

<sup>&</sup>lt;sup>7</sup> For users or other persons, this definition is restricted to events related to the investigational product.

<sup>8</sup> The term "life threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe. (Source: ICH E2A clinical safety data management: definitions and standards for expedited reporting).

<sup>&</sup>lt;sup>9</sup> Planned hospitalization for a pre existing condition, or a procedure required by the CSP, without serious deterioration in health, is not considered a SAE. (Source: ISO14155:2011).

Print date:

2022-07-26 17:40

Exceptions from AE reporting are normal fluctuations in pre-existing diseases. However, pre-existing illnesses that deteriorates (in intensity or frequency) shall be reported as AEs.

When an AE is related to a device deficiency (refer to section 7.8), including technical device malfunction, the AE shall be recorded on the AE form in the eCRF and the technical complaint shall be reported separately on the clinical study complaint form.

Investigators, or other study site personnel, shall record all AEs in the eCRF, including:

- a) Event term (recorded in standard medical terminology and avoiding abbreviations)
- b) Description of event and affected area
- c) Start date (first day with symptoms)
- d) Stop date (last day with symptoms)
- e) Intensity (mild, moderate, or severe according to definition in Section 7.7.3.1)
- f) Seriousness (serious or not serious, according to definition in Section 7.7.3.2)
- g) Causal relationship to study product or study product injection procedure (yes or no)
- h) Action taken (none, medication treatment, non-medication treatment, or other procedures/tests, subject withdrawn)
- i) Outcome of the AE (ongoing, recovered, recovered with sequelae, death, chronic/stable, not recovered at the end of the study)

The pre-defined, expected post-treatment events shall be assessed separately. These event shall be collected daily by subjects in a Diary for up to 28 days after each treatment.

#### 7.7.3.1 *Intensity*

Intensity will be recorded for each reported AE. The following definitions of intensity are to be used:

Mild: Awareness of symptoms or signs, but easily tolerated (acceptable)

**Moderate:** Enough discomfort to interfere with usual activity (disturbing)

**Severe:** Incapacity to work or to do usual activity (unacceptable)

If the intensity changes within one day, the maximum intensity of the AE during that day shall be recorded.

#### 7.7.3.2 *Causal relationship and seriousness*

Each AE, serious as well as non-serious, shall be assessed by the Investigator for causal relationship with the study product and its use (the injection procedure) and for seriousness (Yes or No) of the event.

A two-point scale (Yes or No response) shall be used for the causality assessments. The Investigators shall be asked to indicate a response to each of the following questions in the eCRF:

- "Do you consider that there is a reasonable possibility that the event may have been caused by the study product?", and
- "Do you consider that there is a reasonable possibility that the event may have been caused by the study product injection procedure?"

Print date:

2022-07-26 17:40

If any of these questions is answered "Yes", the AE is considered related.

Each AE will also be assessed for causal relationship and seriousness by the Sponsor, in order to fulfil regulatory requirements.

### 7.7.4 Reporting of adverse events

Adverse event reporting on each subject shall start upon enrollment (i.e. randomized and/or treated) in the study. Any events that occur after the subject signs the ICF but before enrollment will be recorded in the subject's medical history.

The reporting shall continue during each follow-up visit (including any telephone contacts and extra visits between planned visits) until the last scheduled visit in the study.

All AEs, non-serious as well as serious, are to be reported as an AE in the eCRF.



### 7.7.6 Reporting of serious adverse events

The Investigator shall report any **SAE** to the CRO **immediately but not later than 24 hours of awareness of the event**. This initial report can be made via e-mail.

In case of difficulty to obtain all the required information within 24 hours, an initial report can be submitted, with the following information as a minimum, irrespective of whether some of it is regarded as preliminary:



Doc id

2022-07-26 17:40

Effective date: 2019-02-21 18:33



The SAE form must be signed and dated by the Investigator. If the initial 24-hour SAE report does not contain full information or if it is made without using the SAE form the fully completed and signed SAE form shall be e-mailed as noted above. A copy of the fully completed SAE form shall be kept at the site.

In addition, the Investigator shall report SAEs to the responsible IRB without undue delay, if applicable according to national regulations. The Investigator is responsible for checking what reporting procedures are applicable for his/her IRB regarding SAEs and final report of the outcome of the study and to comply with such reporting procedures during the study period. For non-urgent complementary information not possible to send by e-mail or fax, please use surface mail.



Doc id 43USSA1705 Sculptra Clinical Study Protocol GALDERMA MA-37876

Print date:

2022-07-26 17:40



#### 7.7.9 Pregnancy

Pregnancy itself is not regarded as an AE.

If there is a pregnancy after the subject has been treated, the subject must continue to be followed and the outcome of pregnancy must be reported even if the delivery occurs after study completion. Additional treatment with study product is not allowed once a pregnancy is noted.

A pregnancy confirmed during the study period after treatment must be reported by the Investigator on a pregnancy report form immediately upon acknowledgement and submitted to the CRO according to contact details specified in section 7.7.6. The report can be prospective or retrospective. Follow-up should be conducted to obtain outcome information on all prospective reports.

Cases that led to fetal distress, fetal death or a congenital abnormality or birth defect are to be regarded as SAEs and shall be reported on the exposure in utero report form to the CRO immediately but no later than 24 hours after the Investigator's awareness. These events shall be handled as SAEs during data processing. Other complications during the pregnancy that are related to the pregnant woman and fulfils any serious criteria, such as pre-eclampsia requiring hospitalization, shall be reported and handled as SAEs. Elective abortions without complications shall not be reported as AEs.

Print date:

2022-07-26 17:40



#### 7.8 Device deficiencies

### 7.8.1 Definition of a device deficiency

A device deficiency is defined as an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety<sup>10</sup>, or performance.

Note: Device deficiencies include malfunctions, use errors, and inadequate labelling.

#### 7.8.2 Recording instructions

When a device deficiency is discovered, Part A of the clinical study complaint form shall be completed by the Investigator or qualified designee and entered into the eCRF. The type of complaint shall be described and injury to the subject or user or unintended exposure to study product shall be reported as applicable. If an injury has occurred, an AE or an SAE form shall be completed as applicable (refer to Section 7.7). If no SAE was experienced as a result of the device deficiency, the Investigator shall assess whether or not the device deficiency could have led to an SAE if:

- Suitable action had not been taken,
- Intervention had not been made or,
- Circumstances had been less fortunate

In Part B of the clinical study complaint form, the Sponsor will make the same assessment.



A device deficiency that led to a SAE and any device deficiency that could have led to a SAE shall be reported to the CRO within 24 hours after the Investigator's awareness (for contact information, see Section 7.7.6).

In order to fulfil regulatory reporting requirements, all deficiencies with the study product must be assessed by both the Investigator and the Sponsor to determine if it could have led to an SAE.

<sup>&</sup>lt;sup>10</sup> Inadequacy of device safety refers to properties of the device which could have or have led to an AE.



If an SAE has resulted from a device deficiency or if either the Investigator or the Sponsor assesses that the device deficiency could have led to a SAE, the sponsor is responsible for reporting the device deficiency to RA and the PI is responsible for reporting it to the IRB.

The deficient study product shall be kept by the study site until the Sponsor has confirmed whether the product shall be returned to Sponsor for further study or if it can be destroyed at the study site.

#### 8. Effectiveness Assessments



Doc id 43USSA1705 Sculptra Clinical Study Protocol GALDERMA MA-37876







sed

Print date:

2022-07-26 17:40



## 9 Data Handling and Management

#### 9.1 Data management

Data management based on GCP refers to the activities defined to achieve safe routines to enter clinical data information into a database, efficiently and avoiding errors. The data management routine includes procedures for handling eCRFs database set-up and management, data entry and verification, data validation, and documentation of the performed activities including information of discrepancies in the process. The data management process will be described in detail in the data management plan (DMP).

The database, the data entry screens and program will be designed in accordance with the CIP and the eCRF. Data validation will be performed by computerized logical checks and manual review. Drugs and events will be coded in accordance with World Health Organization (WHO) Drug and medical dictionary for regulatory activities (MedDRA) dictionaries as specified in the DMP. SAEs in the clinical database will be reconciled against the data in the safety database.

When all efforts have been made to ensure that the data recorded in the eCRFs and entered in the database is as correct and complete as possible, the clinical database will be locked. Study data will be transferred to SAS datasets, which thereafter will be write-protected. Statistical analyses will be generated in SAS using data from the locked datasets.

#### 9.2 Electronic case report forms

A 21 Code of Federal Regulations Part 11-complaint electronic data capture application will be used to collect, modify, maintain, archive, retrieve, and transmit study data. An eCRF is required and shall be completed electronically for each screened subject (screening visit) and enrolled subjects (subsequent visits).

The eCRF includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Study data shall be entered directly from the source documents, which are to be defined at each site before inclusion of the first subject.

Authorized study site personnel designated by the Investigator shall complete data collection. Appropriate training and security measures shall be completed with all authorized investigation site personnel prior to the study being initiated and any data being entered into the system for any subject.

The study data is the sole property of the Sponsor and shall not be made available in any form to third parties, except for authorized representatives of appropriate RA, without written permission from the Sponsor. At the end of the study, electronic data are kept at the Sponsor and a copy (provided by the vendor) at the study site as part of the Investigator file.

Any delegation of collection of data shall be specified in a signature and delegation log.

Print date:

2022-07-26 17:40

#### 9.2.1 Data entry

All data shall be entered in English. The eCRFs should always reflect the latest observations on the subjects participating in the study. Therefore, every efforts should be made to complete the eCRFs within a reasonable time frame after the subject's visit. The subject's identity must always remain confidential, i.e. the name and address of the subjects must not be registered in the eCRFs or in the database. The Investigator must verify that all data entries in the eCRFs are accurate and correct. If some assessments are not done, or if certain information is not available, not applicable or unknown, the Investigator shall indicate this in the eCRF. The Investigator shall electronically sign off the study data. By signing, the Investigator takes responsibility for the accuracy, completeness, and legibility of the data reported to the Sponsor in the eCRF.

#### 9.2.2 The query process

The monitor shall review the eCRFs and evaluate them for completeness and consistency. Each eCRF shall be compared with the respective source documents to ensure that there are no discrepancies between critical data. All entries, corrections, and alterations shall be made by the PI or his/her authorized designee. The monitor cannot enter data in the eCRFs. Once study data have been submitted to the central server via the eCRF, corrections to the data fields will be audit trailed, meaning that the reason for change, the name of the person who made the change, together with time and date will be logged. Roles and rights of the site personnel responsible for entering study data into the eCRF shall be determined in advance. If discrepant data is detected during review of the data, either by the Sponsor or by its representatives, the responsible data manager or monitor shall raise a query in the electronic data capture application. The query shall state the question or data to be changed and shall be resolved in the system by the PI or his/her authorized designee. The appropriate study site personnel shall answer the queries in the eCRF within a reasonable timeframe Answered queries will be audit trailed by the electronic data capture application meaning that the name of study site personnel, time, and date is logged. Answered queries will then be closed by the appropriate study personnel (i.e. data manager, site monitor, etc.)

#### 9.2.3 User identification

eCRF records will be automatically appended with the identification of the creator, by means of their unique User ID. Specified records shall be electronically signed by the Investigator to document his/her review of the data and acknowledgement that the data are accurate. This will be facilitated by means of the Investigator's unique User ID and password; date and time stamps will be added automatically at time of electronic signature. If an entry in an eCRF requires change, the correction shall be made in accordance with the relevant software procedures.

#### 9.2.4 Audit trail

All changes will be fully recorded in a protected audit trail and a reason for the change shall be stated. Once all data have been entered, verified, and validated, the database will be locked.

#### 9.3 Source documents

Source documents are all documents used by the Investigator or hospital that relate to the subject's medical history, that verifies the existence of the subject, the inclusion and



2022-07-26 17:40

exclusion criteria, and all records covering the subject's participation in the study. They include laboratory notes, memoranda, material dispensing records, subject files, etc.

The Investigator is responsible for maintaining source documents. These shall be made available for inspection by the monitor at each monitoring visit. The Investigator must submit a completed eCRF for each subject for whom signed informed consent has been collected. All supportive documentation submitted with the eCRF, such as laboratory or hospital records, shall be clearly identified with the CTN and subject number. Any personal information, including name, shall be removed or rendered illegible to preserve individual confidentiality.

#### 9.4 Record keeping and access to source data

The Investigator/Institution shall permit study-related monitoring, audits, IRB review, and RA inspections and shall provide direct access to the source data/medical record including the identity of all participating subjects (sufficient information to link records, i.e. eCRF, medical records, original signed informed consent forms and detailed records of study product accountability). The records shall be retained by the Investigator as required by local legislation and international guidelines. Any transfer of responsibility for storage of the records shall be documented and the Sponsor shall be informed in writing.

The Sponsor shall verify that each subject has consented in writing to direct access to the original medical record/source data (by the use of written subject information and signed informed consent). The data recorded in the eCRFs will be checked for consistency with the source documents/medical record by the monitor during monitoring (source data verification; SDV). In order to be able to perform SDV, information about each subject's participation in the study has to be detailed in the medical record.

### 9.5 Document and data retention

All records pertaining to the conduct of the study, including signed eCRFs, informed consent forms, study product accountability records, source documents, and other study documentation must be retained for as long as is specified in the CTA. Measures shall be taken to prevent accidental or premature destruction of these documents (e.g. protection against damage and unauthorized access, preferably by storage in a fire-proof cabinet).

It is the Investigator's responsibility to inform the Sponsor in writing if the Investigator file is moved or if the responsibility for the documents is transferred to someone else.

#### 10 Statistical Methods

#### 10.1 General



Print date:

2022-07-26 17:40





## 10.3 Demographics, baseline assessments, and subject characteristics

Demographic endpoints and subject characteristics will be presented using descriptive statistics.

## 10.4 Primary effectiveness analysis



Doc id 43USSA1705 Sculptra Clinical Study Protocol GALDERMA MA-37876

Print date:

2022-07-26 17:40

### 10.5 Secondary effectiveness analysis

Exact confidence intervals will be used for the proportions, i.e. they will be based on the binomial distribution.



#### 10.6 Safety analysis

Number and percentage of subjects reporting each pre-defined, expected, post-treatment symptoms, as collected in the 28-day diary, will be presented in total and by maximum severity.

All AEs will be coded according to MedDRA and summarized by system organ class (SOC), preferred term (PT) and treatment.



Doc id 43USSA1705 Sculptra Clinical Study Protocol GALDERMA MA-37876

Print date:

2022-07-26 17:40



#### 10.7 Subgroup analyses



### 10.8 Handling of missing data

Number of missing values will be summarized and reported as appropriate.

For ITT analysis of the primary endpoint, missing values will be imputed using the baseline observation carried forward (BOCF) method.

### 10.9 Interim analysis

Since the Sponsor is not blinded to treatment in this study, available data may be analyzed prior to study completion.

#### 10.10 Withdrawals and deviations

All withdrawn subjects will be listed individually, including at least subject number, date and reason for withdrawal, and last visit performed.

Subjects with CIP deviations will be listed individually, including subject number and observed deviation. Depending on the seriousness of the deviation, subject might be excluded from the PP population, which shall be documented prior to database lock.

Deviations from the statistical plan will be documented in the statistical report.

#### 10.11 Sample size



Print date:

2022-07-26 17:40



## 11 Protection of personal data

All processing of personal data must be carried out in accordance with national legislation concerning the protection of personal data. The Institution and the Investigator are responsible for complying with all requirements pursuant to national legislation in which the Institution and the Investigator are located. The Sponsor will ensure that all requirements for data processing are fulfilled.

The Investigator understands that clinical studies conducted under an IDE are exempt from the study subject identifier confidentiality provisions of the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and the study subject should be made aware of this exception in the informed consent. The Institution and Investigator are jointly responsible for providing sufficient information to all subjects to enable them to give their informed consent not only to the participation in the investigation, but also to the processing of Personal Data. Such information includes information regarding the purposes of the processing, the length of time during which Personal Data will be stored, the right of access to stored Personal Data and the right to correction or purging of incorrect or obsolete Personal Data. A subject may also withdraw his or her consent at any time.

A subject who withdraws his or her consent to the processing of Personal Data must be considered to have withdrawn from the investigation but the data collected until the consent was withdrawn may be used in the statistical analyses.

Authorized representatives from the Sponsor or a RA may visit the investigational site to perform audits/inspections, including source data verification, i.e., comparing data in the subjects' medical records and the eCRF. Data and information will be handled with strict confidentiality.

The study shall include collection and processing of personal data as specified in the Regulation (EU) 2016/679 (General Data Protection Regulation, GDPR) on the protection of individuals with regard to the processing of personal data. For the purposes of the study, Sponsor will be considered the data controller, and Institution and PI will both be considered data processors.

## 12 Quality Control and Quality Assurance

#### 12.1 Quality control



2022-07-26 17:40

On-site monitoring of the study will be arranged by the Sponsor according to GCP guidelines to verify that the rights and well-being of the subjects are protected, the reported data are accurate, complete, verifiable from source documents, and that the conduct of the study complies with the approved CIP, subsequent amendment(s), GCP and the applicable regulatory requirements.

Any CIP deviation shall be reported in the eCRF, which will be verified, discussed, and collected by the monitor and appropriate actions will be taken. The Investigator is responsible for promptly reporting any deviations from the CIP that affects the rights, safety or well-being of the subject or the scientific integrity of the study, including those that occur under emergency circumstances, to the Sponsor as well as the IRB if required by national regulations. Deviations will be reviewed to determine the need to amend the CIP or to terminate the study. Handling of CIP deviations will be performed as described in the monitoring manual.

#### 12.2 Quality assurance

The study site may be subject to quality assurance audit by the Sponsor as well as inspection by appropriate RA. It is important that the Investigator and other relevant study site personnel are available during the monitoring visits, possible audits, and inspections, and that sufficient time is devoted to the monitoring process.

Each participating member of the study site team shall provide a curriculum vitae (CV) or equivalent that demonstrates their qualifications to conduct the study.

It is the responsibility of the Investigator to ensure that all personnel involved in the study are fully informed of all relevant aspects of the study, including detailed knowledge of and training in all procedures to be followed. All Investigators and other responsible persons shall be listed together with their function in the study on the signature and delegation log.

#### 12.3 Changes to the clinical study protocol

The Investigator and other site personnel involved in the study must not implement any deviation from or changes to the CIP without agreement with the Sponsor and prior review and documented approval from the IRB except where necessary to eliminate an immediate hazard to the subjects. All changes to the final CIP must be documented in a written protocol amendment. However, administrative changes are to be documented in the Sponsor file without requiring a protocol amendment. The Sponsor will assess if the changes require prior FDA approval, and inform the Investigator when such approval has been received.

## 13 Financing, Indemnification, and Insurance

The CTA outlines the compensation and payment terms of the study. The CTA must be signed before the first subject is screened in the study. If there are differences between the CTA and the CIP regarding certain rights and obligations, the CTA is the prevailing document. The Sponsor's obligations in this clinical study are covered by Galderma's global general liability program. An insurance certificate will be provided upon request. The Institution/Investigator is obligated to maintain insurance coverage for their obligations in the clinical study according to the CTA.

## 14 Publication Policy

The Investigator's, Institution's, and Sponsor's obligations regarding intellectual property

Print date:

2022-07-26 17:40

rights, confidentiality, and publications are described in detail in the CTA.

This study will be displayed on clinicaltrials.gov in accordance with local regulations. The aim is to submit the results of this study for publication. Everyone who is to be listed as an author of the publication shall have made a substantial, direct, intellectual contribution to the work. Authorship will be based on (1) substantial contributions to the conception or design of the work; or the acquisition, analysis, or interpretation of data for the work; and (2) drafting the work or revising it critically for important intellectual content; and (3) final approval of the version to be published; and (4) agreement to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved<sup>12</sup>. Conditions 1, 2, 3, and 4 must all be met in order to be designated as author. Those who do not meet all four criteria will be acknowledged. Among the authors that fulfil the above mentioned criteria, one author will be appointed by to take primary responsibility for the overall work as primary author.

### 15 Suspension or Premature Termination

The Sponsor will suspend or terminate the study when so instructed by the IRB or FDA, or if it is judged that the subjects are subjected to unreasonable risks, or for valid scientific or administrative reasons, or for business reasons.

The Sponsor may also decide to close a single study site due to unsatisfactory subject enrollment or non-compliance with the CIP, GCP, or applicable regulatory requirements.

In the event of premature termination, the Sponsor will provide information on the handling of currently enrolled subjects who have not completed the study.

<sup>&</sup>lt;sup>12</sup>Defining the role of authors and contributors, compiled by the International Committee of Medical Journal Editors (ICMJE) (http://www.icmje.org).

Print date:

2022-07-26 17:40

### 16 References

- https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medicalresearch-involving-human-subjects/
- 2. <a href="https://www.verywell.com/fitzpatrick-classification-scale-1069226">https://www.verywell.com/fitzpatrick-classification-scale-1069226</a>
- 3. Alessio R, Rzany B, Eve L, et al. European expert recommendations on the use of injectable poly-L-lactic acid for facial rejuvenation. *Journal of Drugs in Dermatology*. 2014; 13(9) P. 1057-1066.
- Fitzpatrick T.B. (1988). The validity and practicality of sun reactive skin types I through VI. Arch. Dermatol. 124, 869–871.
- 5. Lemperle, G. A Classification of Facial Wrinkles. Plastic Reconstructive Surgery. 2001: 1735-1750.
- Lorenc P, Greene T, Gottschalk RW. Injectable Poly-L-Lactic Acid: Understanding its use in the current era. J Drugs Dermatol. 2016; 15(6) P. 759-762.
- Rossner F, Rossner M, Hartmann V, et al. Decrease of reported adverse events to injectable polylactic acid after recommending an increased dilution: 8-year results from the Injectable Filler Safety study. J Cosmet Dermatol. 2009; 8(1) P. 14-18.
- Sculptra® Aesthetic Instructions for Use. Galderma Laboratories L.P., Fort Worth Texas, USA (07/2016).
- Vleggaar D, Fitzgerald R, Lorenc ZP, et al. Consensus recommendations on the use of injectable poly-L-lactic acid for facial and nonfacial volumization. *J Drugs Dermatol*. 2014; 13 (4) P. 44-50.
- Vleggaar D, Fitzgerald R, Lorenc P. The history behind the use of injectable poly-L-lactic acid for facial and nonfacial volumization: the positive impact of evolving methodology. *J Drugs Dermatol*.2014; 13(4) P.32-34.
- Vleggaar D, Fitzgerald R, Lorenc ZP. Understanding, avoiding, and treating potential adverse events following the use of injectable poly-L-lactic acid for facial and nonfacial volumization. *JDrugs Dermatol*. 2014;13(4) P.35-39.

9.



# 17 Appendices





Effective date: 2019-02-21 18:33

43USSA1705 Sculptra Clinical Study Protocol

Doc id

Print date:

MA-37876

2022-07-26 17:40

Appendix 2



Title
43USSA1705 Sculptra Clinical Study Protocol

Doc id

Print date:

MA-37876

2022-07-26 17:40

Appendix 3.



Print date: 2022-07-26 17:40

GALDERMA
Title
43USSA1705 Sculptra Clinical Study Protocol

MA-37876

Effective date: 2019-02-21 18:33



Print date: 2022-07-26 17:40

GALDERMA

Title

43USSA1705 Sculptra Clinical Study Protocol

MA-37876

Effective date: 2019-02-21 18:33



43USSA1705 Sculptra Clinical Study Protocol Doc id ♣ GALDERMA MA-37876

Print date:

2022-07-26 17:40

